CLINICAL TRIAL: NCT00470990
Title: Effect of Varying Testosterone Levels on Insulin Sensitivity in Normal and IHH Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: American Diabetes Association (Other)
Responsible Party: Frances J. Hayes, MD, Massachusetts General Hospital, Boston MA
Model: Crossover | Masking: None
Other Study IDs: 2002-P-001445 (completed)
Record Dates: First submitted 2007-05-07; First posted 2007-05-08 (Estimated); Last update posted 2011-04-20 (Estimated); Status verified 2011-04

CONDITIONS: Hypogonadism
Keywords: IHH; Kallmann syndrome; hypogonadism
MeSH Terms: conditions — Hypogonadism; Kallmann Syndrome | interventions — acyline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: GnRH antagonist (Acyline) — 3 Subcutaneous injections (300 mcg/kg) over 36 days
  Other Names: IND # 62,621

SUMMARY:
Type 2 diabetes is one of the most common metabolic disorders in the U.S, estimated to affect 16 million Americans. Established risk factors for this disease include obesity, increased waist/hip ratio, high insulin levels in the blood, and insulin resistance. Testosterone may play a role in developing or preventing diabetes, but we do not yet know for sure. The purpose of this research study is to determine if changing testosterone levels in men will result in changes in insulin sensitivity. Information learned form this research study may have important public health implications and may point to new strategies for treating or preventing diabetes.

DETAILED DESCRIPTION:
The overall aim of this study is to examine the effect of testosterone on insulin sensitivity using the models of acute and chronic hypogonadism. All subjects will be in good general health and 2 groups of men will be studied in this protocol:

1. Thirty healthy normal men aged 18-75 years with normal blood pressure, normal testosterone levels, and not taking any medications known to influence glucose homeostasis or testosterone
2. Ten adult men (over the age of 18) with idiopathic hypogonadotropic hypogonadism (IHH)and normal thyroid, adrenal, and growth hormone axes as well as normal prolactin levels and no abnormalities on imaging of the hypothalamic-pituitary region. These men will be on no medications known to influence glucose homeostasis and will have been off hormone therapy for a suitable washout period depending on the type of prior androgen replacement.

ELIGIBILITY:
Inclusion Criteria:

Healthy men:

Good general health,

* Normotensive,
* Normal testosterone levels,
* No medications known to influence glucose homeostasis or testosterone levels

IHH men:

* Good general health;
* Normal thyroid, adrenal, and GH axes;
* Normal prolactin levels;
* No abnormalities on imaging of the hypothalamic-pituitary region;
* No medications known to influence glucose homeostasis;
* Must have been off hormone therapy for a suitable washout period depending on the type of prior androgen replacement

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2002-10; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
insulin sensitivity | 2 timepoints: with a normal serum testsoterone and in a castrate state of low serum testoserone

SECONDARY OUTCOMES:
body composition | 2 timepoints: with a normal serum testsoterone and in a castrate state of low serum testoserone

CONTACTS AND LOCATIONS:
Overall Officials: Frances J Hayes, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States